CLINICAL TRIAL: NCT04602702
Title: INVESTIGATING THE POTENTIAL OF SHORT-TERM PATIENT DERIVED XENOGRAFTS FOR PERSONALIZED MEDICINE FOR PATIENTS WITH METASTATIC SOLID TUMORS: A Non-interventional Clinical Trial.
Brief Title: Hyper-Personalized Medicine Using Patient Derived Xenografts (PDXovo) for Metastatic Solid Tumors
Acronym: PDXovo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: SUN-2047
Record Dates: First submitted 2020-09-10; First posted 2020-10-26 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Kidney Neoplasm; Carcinoma, Renal Cell; Metastatic Solid Tumor
Keywords: hyper-personalized medicine; patient derived xenograft; chick embryo
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — metastasectomy specimens, needle core biopsies, thoracentesis, paracentesis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Investigators will use novel PDX (patient-derived xenograft) technology to form xenografts using material from metastatic solid tumor patients. Xenografts will be treated with a panel of drugs to determine which agent(s) yield the greatest anti-tumor effect on the xenograft.

DETAILED DESCRIPTION:
The goal is to use PDXovos, which are chick embryos cultivated in an ex ovo fashion that will act as a xenograft host, for drug paneling. Chick embryos as a PDX host model system offer multiple advantages, such as increased tumor take rates, rapid drug testing, a short evaluation timeframe, and an undeveloped adaptive immune system. Collectively, these advantages allow for implantation of tumor xenografts, subsequent growth in vivo, subsequent drug challenge, and subsequent evaluation for anti-tumor effects.

Patients with metastatic forms of solid tumors will be enrolled regardless of subtype. Metastases will be provided either via metastasectomy or needle core biopsy of metastatic deposits. Spinal and intracranial metastases will be included. Thoracentesis and paracentesis fluid samples yielding tumor tissue will also be included.

Tissue will be processed and briefly cultured in vitro. Upon authentication and expansion to a suitable number of cells, xenografts will be formed in the chick embryo pre-clinical model. After implantation (2 days later), drug treatments will be applied topically to each xenograft's surface. Drug treatments are: sunitinib, pazopanib, axitinib, temsirolimus, cabozantinib, gemcitabine (N>18/treatment group).

Evaluation of xenografts for anti-tumor effects will be performed via ultrasound imaging (changes in tumor volume and tumor vascularity) and confirmed by histology (H&E, TUNEL, CD31+ microvessel density). Treatments will be compared to vehicle control (5% DMSO in saline) treated xenografts. ANOVA (2-way, p<0.01, bon ferroni alpha corrected) analysis will be performed to identify treatments that lead to the greatest decrease in tumor volume and tumor vascularity (ultrasound imaging metrics). Agents identified will not be used to intervene in clinical care. Objective response rates with clinically chosen drug in each patient will be compared to the corresponding PDX drug panel results using kappa analysis.

ELIGIBILITY:
Patient eligibility:

Localized solid tumor inclusion criteria:

i) Age 18+ ii) localized solid tumor irrespective of subtype undergoing curative surgery iii) Consent to provide tumor tissue for this research

Metastatic cancer inclusion criteria:

i) Age 18+ ii) metastatic cancer irrespective of subtype undergoing a needle biopsy or resection of lung, liver or brain as part of their routine clinical care.

iii) metastatic cancer irrespective of disease site undergoing a thoracentesis or paracentesis as part of their routine clinical care.

iv) measurable disease as per RECIST 1.1 criteria v) Consent to provide tumor tissue for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic solid tumors identified at Sunnybrook Health Sciences Centre - Odette Cancer Centre
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response | 3-9 months
  Complete Response, Partial Response
Stable Disease Response | 3-9 months
Progressive Disease Response | 3-9 months

CONTACTS AND LOCATIONS:
Overall Officials: Georg Bjarnason, MD, Principal Investigator — Sunnybrook Hospital/Odette Cancer Centre; Elyse Watkins, BSc, PGDip, Study Director — Sunnybrook Hospital/Odette Cancer Centre; Nir Lipsman, MD, Principal Investigator — Sunnybrook Hospital
Locations (1):
- Odette Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No